CLINICAL TRIAL: NCT00421135
Title: A Protocol for the Safety and Tolerance of Intravenous Isophosphoramide Mustard (IPM) in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Jonathan Lewis, MD PhD Chief Medical Officer, ZIOPHARM Oncology, Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPM1001
Record Dates: First submitted 2007-01-10; First posted 2007-01-11 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — palifosfamide lysine

ARMS (1):
- Single Arm (Experimental): ZIO-201
  Interventions: Drug: ZIO-201

INTERVENTIONS:
Drug: ZIO-201 — ZIO-201 as a single dose given once every 21 days. This is a dose escalation arm.

SUMMARY:
The study of safety of Isophosphoramide Mustard (IPM) in the treatment of advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic and /or unresectable disease state after previous standard chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-02; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
toxicities | 6 months

SECONDARY OUTCOMES:
pharmacokinetics | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Lewis, MD, PhD, Study Director — ZIOPHARM Oncology, Inc
Locations (2):
- United States (2):
  - Santa Monica, California
  - Detroit, Michigan